CLINICAL TRIAL: NCT02639403
Title: Palliative Short-Course Radiotherapy in Rectal Cancer: A Phase II Study
Brief Title: Palliative Short-Course Radiotherapy in Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Rectal Neoplasms
Keywords: Rectal cancer; Radiotherapy; Occlusion
MeSH Terms: conditions — Rectal Neoplasms; Bites and Stings | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RT for Obstructing Rectal Cancer (Experimental): Conformal three-dimensional RT was planned (3D-RT) in patients with obstructing rectal cancer not amenable for curative resection
  Interventions: Radiation: Conformal three-dimensional Radiotherapy

INTERVENTIONS:
Radiation: Conformal three-dimensional Radiotherapy — Conformal three-dimensional RT was planned (3D-RT) using the Oncentra-Masterplan treatment planning system (Nucletron B.V., Veenendaal, Netherland). Short course RT (total, 25 Gy; 5 fraction in 5 days) will be delivered with an isocentric four-field box technique.

SUMMARY:
Radiotherapy (RT) is a potentially effective method in the treatment of symptoms of rectal carcinomas. Nevertheless, almost all the evidences about palliative RT in rectal cancer have been published more than two decades ago and were based on 2D conventional RT, which is nowadays no longer used. Consequently, prospective studies on the efficacy of 3D-RT in the management of symptomatic rectal cancer are still lacking. The aim of this prospective study was to assess the efficacy of palliative short-course 3D RT (SCRT) in patients with symptomatic obstructive rectal cancer.

DETAILED DESCRIPTION:
Colorectal carcinoma is one of the cancers with higher incidence, although a progressive decrease in both incidence and mortality rates has been recently recorded in European countries. Rectal cancer may be diagnosed when the disease is at an advanced stage, causing obstructing symptoms. Colostomy represents a standard treatment option in these patients although it negatively impacts on quality of life. Consequently, alternative treatments have been proposed such as self-expandable metallic stent or thermal ablative treatments (i.e. laser or argon plasma coagulation endoscopic treatments), which are, however, not complication-free and not always feasible.

Radiotherapy (RT) is a potentially effective method in the treatment of symptoms of rectal carcinomas. Nevertheless, almost all the evidences about palliative RT in rectal cancer have been published more than two decades ago and were based on 2D conventional RT, which is nowadays no longer used. Consequently, prospective studies on the efficacy of 3D-RT in the management of symptomatic rectal cancer are still lacking.

The aim of this prospective study was to assess the efficacy of palliative short-course 3D RT (SCRT) in patients with symptomatic obstructive rectal cancer. This trial was a prospective Phase II study performed at the Fondazione di Ricerca e Cura "Giovanni Paolo II" in Campobasso (Italy).

Therapy Radiotherapy During the simulation process, patients were immobilized in prone position on an up-down table, a device aimed at reducing small-bowel irradiation. To limit the organ motion, patients were instructed to empty the bladder and drink 300 cm3 of water one hour before CT-simulation and before every daily treatment fraction. After oral administration of contrast medium to allow bowel localization, simulation CT images were taken in 5 mm increments over the region of interest. Delineation of the clinical target volume 1 (CTV1) included the gross tumor volume (GTV, both primary tumor and enlarged pelvic nodes) and the corresponding mesorectum plus 2 cm cranio-caudally. The planning target volume (PTV) was the CTV plus 0.8 cm margin in all directions. Organs at risk (OARs) were contoured as follows: 1) the small intestine was defined as all intestinal loops below the sacral promontory (recto-sigmoid junction excluded); 2) femoral heads were contoured from the cranial extremity to the level of the lower margin of ischial tuberosities; 3) the bladder was contoured entirely with no distinction between the wall and its content. Conformal three-dimensional RT was planned (3D-RT) using the Oncentra-Masterplan treatment planning system (Nucletron B.V., Veenendaal, Netherland). Short course RT (total, 25 Gy; 5 fraction in 5 days) was delivered with an isocentric four-field box technique. Dose was specified according to the ICRU Report 62. Dose-volume histograms (DVHs) were calculated for the PTV and OARs and the QUANTEC constraints were followed. Radiotherapy was delivered by 10-15 MV photon energy. The beams were delivered by an Elekta Precise Linac (Elekta Oncology Systems, Crawley, UK) equipped with standard multi leaf collimators (MLC). A daily online correction protocol of isocenter position was applied using portal imaging, with set-up correction in case of deviations > 0.5 cm in any direction. All stages of the treatment planning process were subjected to a systematic independent check procedure, as previously described. In patients with grade 3-4 toxicity, RT was suspended and treatment was resumed after recovery from toxicity in the degree ≤ 2.

Chemotherapy Use of chemotherapy was allowed based on the referring physician preferences, comorbidities and age. Chemotherapy was discontinued during RT, one week before and after the delivery of RT.

Statistical Analysis Primary end-point of the present study was the rate of complete response (CR) of obstructive symptoms following radiation treatment. According to the Simon's optimal design, the study required the enrollment of 9+8 patients in order to detect a significant rate of CR of obstructive symptoms (error probability limits: alpha 0.05; beta 0.2). In case of no detection of CR of obstructive symptoms in the first 9 enrolled patients, the interruption of enrollment and the closure of the study were planned. In case of detection of at least 1 CR of obstructive symptoms the study design required the recruitment of at least 8 additional patients for the final evaluation of symptoms response rate. To account for a possible non-participation rate of 5%, we increased the sample size of the second stage to nine subjects. Continuous variables were reported as median with range. Categorical variables were reported as proportion and percentage. The survival curves were computed with the Kaplan-Meier method. Statistical analysis was performed with SPSS v. 22 (IBM Corp., Armonk, NY, US) and Stata 14.1 SE (Stata corporation, College Station, TX, US)

ELIGIBILITY:
Inclusion Criteria:

* (i) rectal adenocarcinoma with obstructive symptoms not amenable for curative treatment due to synchronous metastases or patient inoperable due to age and/or comorbidities;
* (ii) symptoms of colorectal obstruction (progressive constipation with abdominal pain arising from less than 2 months, vomiting and/or diarrhea) and/or signs of obstruction at radiological examinations (presence of air-fluid levels or the presence of distended colon upstream neoplastic stenosis of the rectum);
* (iii) candidates for derivative colostomy;
* (iv) bi-dimensionally measurable disease;
* (v) Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
* (vi) able to provide a written informed consent.

Exclusion Criteria:

* (i) RT within 6 months in the same anatomical area before the initiation of study treatment;
* (ii) clinically detectable ascites;
* (iii) pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change of the obstructive symptoms | Clinical evaluation was performed before commencement of RT, 4 weeks after the end of treatment and every 6 months until the established length of follow up (3 years) or death.

SECONDARY OUTCOMES:
Change of the overall symptoms | Before commencement of RT, 4 weeks after the end of treatment and every 6 months until the established length of follow up (3 years) or death.
Change of the tumor mass volume | Before commencement of RT, 4 weeks after the end of treatment and every 6 months until the established length of follow up (3 years) or death.
Number of participants with treatment-related adverse events as assessed by National Cancer Institute Common Toxicity Criteria v4.0 | Before commencement of RT, 4 weeks after the end of treatment and every 6 months until the established length of follow up (3 years) or death.
Overall survival | At the end of follow-up (3 years after RT) or until death of patient
Obstruction/colostomy-free survival | At the end of follow-up (3 years after RT) or until death of patient

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, Professor, Study Director — Policlinico S.Orsola-Malpighi, University of Bologna, Bologna, Italy